CLINICAL TRIAL: NCT01127113
Title: Inflammatory Cell Labelling and Tracking With Magnetic Resonance Imaging After Myocardial Infarction
Brief Title: Inflammatory Cell Trafficking After Myocardial Infarction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EDO001
Record Dates: First submitted 2010-04-13; First posted 2010-05-20 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2014-12

CONDITIONS: Myocardial Infarction; Inflammation
Keywords: Myocardial infarction; Magnetic resonance imaging; Nanoparticles; Mononuclear cells; Cell tracking
MeSH Terms: conditions — Myocardial Infarction; Inflammation | interventions — ferumoxides; Contrast Media

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SPIO-labelled mononuclear cells (Active Comparator)
  Interventions: Other: Infusion of investigational product; Other: Cardiac magnetic resonance imaging
- Unlabelled mononuclear cells (Placebo Comparator)
  Interventions: Other: Infusion of investigational product; Other: Cardiac magnetic resonance imaging
- SPIO alone (Active Comparator)
  Interventions: Other: Infusion of investigational product; Other: Cardiac magnetic resonance imaging

INTERVENTIONS:
Other: Infusion of investigational product — The investigational product will be delivered via intravenous infusion
  Other Names: The investigational product will be either:; 1) Unlabelled autologous mononuclear cells; 2) Endorem (Guerbet, Paris) contrast alone; 3) Autologous mononuclear cells labelled with Endorem
Other: Cardiac magnetic resonance imaging — Cardiac MRI will be performed prior to infusion of investigational product and 1, 2, 7 and 30 days after.

SUMMARY:
Myocardial infarction (heart attack) is usually the consequence of rupture of a fatty 'plaque' in a heart artery. The presence of this fat and debris causes the propagation of a blood clot and blockage of the artery. The heart muscle normally supplied by the artery becomes deprived of oxygen and, if starved for long enough, this area of muscle dies. Much of the heart muscle damage is caused by overactivation of inflammatory cells. Whilst inflammation can be beneficial in healing processes, there is accumulating evidence that overactivation of inflammatory processes contributes to further muscle damage and cell death during myocardial infarction. We have recently developed a means of labelling human blood cells with 'nanoparticles' of iron oxide which can then safely be reinjected into the blood to allow the cells to be tracked and seen in the body using a conventional magnetic resonance scanner.

In the proposed study we aim to recruit patients with recent heart attacks to perform similar cell labelling and reinjection of labelled cells into the same volunteer's blood stream via the arm to track the fate of the blood cells over the course of days to months. We think that the labelled inflammatory cells will 'home' to the site of the heart attack and will be visible using magnetic resonance imaging (MRI) of the heart. We aim not only to highlight the role of inflammatory cells in myocardial infarction, but also propose that, if successful, this technique could be used in the future to assess the effects of antiinflammatory treatments currently being developed for the treatment of patients with heart attacks. The technique could also be extended to allow labelling of other cell types, including stem cells, to let us further understand how these cells may contribute to repair of damaged organs including the heart.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with acute ST segment elevation myocardial infarction:

  * 1 mm ST elevation in at least two contiguous limb leads, or
  * 2 mm ST elevation in at least two contiguous praecordial leads, or new onset bundle branch block
* Successful treatment with primary percutaneous coronary intervention Restoration of TIMI grade 3 flow in infarct-related artery
* Troponin I ≥10 IU/mL at 12 hours after the onset of chest pain
* Age 18 - 80 years

Exclusion Criteria:

* Left main stem or severe multi-vessel coronary artery disease
* Continued symptoms of angina at rest or minimal exertion
* Atrial fibrillation
* Symptomatic heart failure; Killip Class ≥2.
* Hepatic or renal failure (estimated glomerular filtration rate <25 mL/min)
* Terminal illness or malignancy
* Anaemia
* Contraindication to magnetic resonance imaging
* Hepatitis B, hepatitis C, HTLV, HIV or syphilis infection
* Patients at risk of allergy to protamine (fish allergy, infertile men, previous vasectomy)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-01; Primary Completion 2015-11 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in cardiac MRI signal intensity from baseline after administration of labelled vs. unlabelled mononuclear cells. | 90 days

SECONDARY OUTCOMES:
Correlation of myocardial MRI signal intensity change from baseline with markers of systemic inflammation. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, MD, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh, Edinburgh, Midlothian, United Kingdom